CLINICAL TRIAL: NCT03212807
Title: Phase II Study Of Durvalumab In Combination With Lenalidomide In Relapsed/Refractory EBV Associated Subtypes Of DLBCL, Primary CNS Lymphoma And Primary Testicular DLBCL - DuRIANS (Durvalumab Revlimid In Aggressive NHL Subtypes)
Brief Title: Study Of Durvalumab and Lenalidomide In R/R EBV Associated DLBCL Subtypes, Primary CNS And Testicular DLBCL
Acronym: DuRIANS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Hold for Combination Studies using Imids and PD1/PDL1 Compounds
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Center Singapore, Singapore (Unknown); National University Hospital, Singapore (Other); Raffles Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDBCC-LYM-16-02
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: EBV Related Non-Hodgkin's Lymphoma; Primary CNS Lymphoma; Primary Testicular Lymphoma
Keywords: Checkpoint inhibition; PDL1; EBV DLBCL; PCNSL
MeSH Terms: interventions — durvalumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Investigational (Experimental): Durvalumab + Lenalidomide
  Interventions: Drug: Durvalumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Durvalumab — Investigational Medicinal Product
Drug: Lenalidomide — Investigational Medicinal Product

SUMMARY:
PHASE II STUDY OF DURVALUMAB IN COMBINATION WITH LENALIDOMIDE IN RELAPSED/REFRACTORY EBV ASSOCIATED SUBTYPES OF DLBCL, PRIMARY CNS LYMPHOMA AND PRIMARY TESTICULAR DLBCL

Patients with relapsed refractory subtypes of DLBCL who fulfill the inclusion / exclusion criteria will be recruited to this trial and treated in this open label, phase 2 trial with the PDL1 inhibitor Durvalumab and Lenalidomide. The combination treatment will be given from the time of recruitment for 6 months when Lenalidomide will be stopped but Durvalumab will continue for a total of 2 years. Response will be assessed by PET / CT scans as per standard lugano criteria.

DETAILED DESCRIPTION:
This is a multi-center, open-label, phase II study of Durvalumab in combination with Lenalidomide for treatment of relapsed/refractory EBV associated DLBCL subtypes, primary testicular lymphoma and primary CNS lymphoma using a Simon's Two-stage Minimax design. Simon's two-stage Minimax design will be used to investigate if the overall response rate (ORR) is at least 45% against a no-interest ORR of 20%.

In the first stage, 13 patients will be accrued. If there are 2 or fewer responses in these 13 patients, the study will be stopped. Otherwise, 8 additional patients will be accrued for a total of 21 patients.This design yields a type I error rate of 5% and power of 80% when the true response rate is 45%.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be ≥ 21 years of age on the day of signing informed consent
3. Histologically proven relapsed / refractory DLBCL classified under the following WHO Subtypes.

   i, EBV Positive DLBCL (of the elderly and immunosuppression associated) ii, T-cell / histiocyte-rich B-cell lymphoma iii, Plasmablastic lymphoma iv, Gray zone lymphoma v, Primary Mediastinal Large B-Cell Lymphoma vi, Primary CNS Lymphoma (DLBCL) vii, Primary testicular lymphoma The biopsy needs to have been obtained within 3 months of signing informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Patients must have received at least one course (1 - 6 cycles) of Immunochemotherapy for example Rituximab + Chemotherapy (CHOP or CHOP like) and must have relapsed or refractory disease at the time of trial entry.
6. Patients should have been deemed ineligible or failed or refused an autologous stem cell transplant in situations where stem cell transplant is the accepted standard of care. In patients with chemo-refractory DLBCL, even if patient is suitable for ASCT, transplant is extremely unlikely to achieve a response and hence such patients can be recruited after careful consideration by the investigator in discussion with the treating physician.
7. Have measureable disease, defined as at least one lesion that can be accurately measured in at least two dimensions on a CT scan or MRI scan in PCNSL. Minimum measurement must be > 15 mm in the longest diameter by >10 mm in the short axis.
8. Minimum life expectancy of 3 months.
9. Adequate hematological function (unless abnormalities are related to lymphoma infiltration of the bone marrow) within 30 days prior to signing informed consent, including:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
   2. Platelet count ≥ 50 x 109/L
   3. Hemoglobin ≥ 8 g/dL
10. Adequate other organ functions as defined in protocol.
11. Must be able to adhere to study visit schedules and other protocol requirements.
12. Females of childbearing potential must:

    1. Have 2 negative pregnancy tests as verified by a Study Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the patient practices complete abstinence from heterosexual contact.
    2. Either commit to complete abstinence from heterosexual contact or agree to use, and be able to comply with, effective contraception without interruption, 30 days prior to starting study drug, during the study therapy (including dose interruptions), and for 30 days after discontinuation of study therapy.
13. Male patients must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or female of childbearing potential while participating in the study, during dose interruptions and for 30 days after discontinuation of study therapy, even if he has undergone successful vasectomy.
14. All patients must:

    1. Have an understanding that the study drug could have a potential teratogenic risk.
    2. Agree to abstain from donating blood while taking study drug, during dose interruptions and for 30 days after discontinuation of study therapy.
    3. Agree not to share study medication with another person.
    4. Agree to be counseled about pregnancy precautions and risk of fetal exposure.
    5. Females must agree to abstain from breast feeding during the study participation and for 30 days after discontinuation of study therapy.
15. Male subjects should not donate sperm or semen while on the study and during breaks (dose interruptions), and for at least 30 days after the last dose of the study medications.

Exclusion Criteria:

The presence of any of the following will exclude a patient from enrolment:

1. Concomitant use of any other investigational agent or device
2. Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxin, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
3. Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Subjects who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of GVHD).
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. i) Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. ii) If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. iii) Toxicity that has not recovered to ≤ Grade 1 is allowed if it meets the inclusion requirements for laboratory parameters defined in points 8 & 9 under inclusion criteria.

   iv) Patients who have had Intrathecal chemotherapy within 2 weeks of trial entry if it was given at the time of diagnostic lumbar puncture could still be included.
5. Known infection with human immunodeficiency virus (HIV).
6. Patient has known clinically active hepatitis B; carriers of hepatitis B are permitted but need to be on appropriate anti-viral therapy or have regular hepatitis B DNA virus monitored as advised by a Gastroenterologist.
7. Neuropathy > Grade 2.
8. Patients who are at a high risk of a thromboembolic event and are not willing to take venous thromboembolic prophylaxis.
9. Myocardial infarction within 6 months prior to enrolment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
10. Clinically significant active infection needing intravenous systemic therapy or uncontrolled intercurrent illness.
11. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
12. Has evidence of active, non-infectious pneumonitis
13. Pregnant or lactating females.
14. Coexistent second malignancy or history of prior malignancy within the preceding 3 years (excluding non-melanoma skin tumors or in situ carcinoma of the cervix).
15. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.
16. Has received a live vaccine within 30 days prior to first dose.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | at least 6 months of follow up
  Overall response rate (ORR) is defined as the proportion of patients with reduction in tumor burden of at least 50%. ORR will be reported with corresponding 95% confidence intervals using the exact binomial method.

SECONDARY OUTCOMES:
Progression free survival | 12 months
  Progression-free survival (PFS) is defined as the time from enrolment to progression or death due to any cause.
Overall Survival | 2 years
  Overall survival (OS) is defined as the time from registration to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Chandramouli Nagarajan, MD FRCPath, Principal Investigator — Singapore General Hospital
Locations (4):
- Singapore (4):
  - National Cancer Center, Singapore
  - National University Hospital, Singapore
  - Raffles Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No